CLINICAL TRIAL: NCT01231178
Title: Alginate Fibers Effect on Body Weight and Risk Markers for Type 2 Diabetes and Cardiovascular Disease.
Brief Title: The Effect of an Alginate Based Beverage on Weight Loss
Acronym: ALGOBES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Prof. Arne Astrup, MD, Head of Department, Department of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B272; Scientific Ethical Committee (Registry Identifier: H-2-2009-155)
Record Dates: First submitted 2010-04-08; First posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-04

CONDITIONS: Obesity; Type 2 Diabetes; Cardiovascular Disease
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alginate based beverage (Active Comparator)
  Interventions: Dietary Supplement: Alginate beverage
- Control beverage (Placebo Comparator)
  Interventions: Dietary Supplement: Control beverage

INTERVENTIONS:
Dietary Supplement: Alginate beverage — The dosage is 3x500ml daily
  Other Names: Protanal
  Arms: Alginate based beverage
Dietary Supplement: Control beverage — The dosage is 3x500ml daily
  Other Names: Maltodextrin
  Arms: Control beverage

SUMMARY:
The project aims to examine the efficacy of a 12-week intake of alginate based ready to drink supplement on development in body weight and body composition, and risk markers for type-2 diabetes and cardiovascular disease in obese subjects.

DETAILED DESCRIPTION:
The study consists of a parallel RCT with 96 overweight/obese subjects enrolled into two treatment arms: placebo or active for 12 weeks. They will undergo examination at time points 0 and 12 weeks where a DXA scan will be performed to assess body composition and a fasting blood sample will be taken. At time points 0, 2, 4, 6, 8, 10 and 12 weeks their weight and waist circumference and number of test products not consumed will be recorded. In addition all subjects receive dietary counselling during the 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Overweight to obese (BMI 28-45 kg/m2)

Exclusion Criteria:

* Chronic diseases including:liver and kidney disease, including P-Alanine aminotransferase (ALT), P-aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT), creatinine kinase and P-lactate dehydrogenase (LD)> 2.0 times the upper limit of normal (ULN) (measured at the screening at the Department of Human Nutrition)
* systemic infections and metabolic diseases that can interfere with energy balance,
* diabetes or fasting blood glucose concentration> 7.0 mM, cardiovascular disease, systolic blood pressure ≥ 160 and / or a diastolic blood pressure ≥ 100 mmHg, hyperlipidemia (total cholesterol> 6.5 mM and triglycerides> 5.0 mM) (measured by the screening at the Department of Human Nutrition)
* Food allergies
* Psychiatric disorders and any clinical condition that makes the person unfit to participate in the experiment
* Use of dietary supplements (during the experimental period and 3 months before study start)
* Provision of blood for example. of donation or other scientific studies (during the trial and 3 months before study start) and hemoglobin <7.5 mmol / l (measured at the screening at the Department of Human Nutrition)
* Smoking (throughout the trial and 6 months before study start)
* Elite Athletes (> 10 hours strenuous exercise per week, self-reported)
* Women who are pregnant or breastfeeding, and post-menustruelle (self reported)

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 Weeks

SECONDARY OUTCOMES:
Blood pressure | 12 weeks
Risk markers for type 2 diabetes | 12 weeks
Risk markers for cardiovascular disease | 12 Weeks
Body composition | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Prof. MD., Principal Investigator — Department of Human Nutrtion
Locations (1):
- Department of Human Nutrition, Frederiksberg, Copenhagen, Denmark

REFERENCES:
- [Derived] Georg Jensen M, Kristensen M, Astrup A. Effect of alginate supplementation on weight loss in obese subjects completing a 12-wk energy-restricted diet: a randomized controlled trial. Am J Clin Nutr. 2012 Jul;96(1):5-13. doi: 10.3945/ajcn.111.025312. Epub 2012 May 30. PMID 22648709